CLINICAL TRIAL: NCT04778293
Title: Effects of Diacutaneous Fibrolysis on Passive Neuromuscular Response and Mechanosensitivity on Posterior Muscular Chain of Lower Limb in Athletes.
Brief Title: Effects of Diacutaneous Fibrolysis on Passive Neuromuscular Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Aida Cadellans Arróniz, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS-2020-04
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hamstring Contractures

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment will be performed by a blinded evaluator at the baseline, immediately after the technique application and 30 minutes after.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): An experienced physiotherapist in the diacutaneous fibrolysis technique will apply the treatment to the lower limb, previously randomized (random.org), in the following musculature and intermuscular septums: quadratus lumbar, gluteus maixum, biceps femoris and semitendinosus. Intervention procedure will last about 10-15 minutes
  Interventions: Other: Diacutaneous fibrolysis
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Diacutaneous fibrolysis — An experienced physiotherapist in the diacutaneous fibrolysis technique will apply the treatment to the lower limb, previously randomized, in the following musculature and intermuscular septums: quadratus lumbar, gluteus maixum, biceps femoris and semitendinosus. Intervention procedure will last about 10-15 minutes
  Arms: Experimental Group

SUMMARY:
Diacutaneous fibrolysis is a physiotherapeutic instrumental technique, used to treat musculoskeletal conditions causing pain and/or movement restriction . It is applied by means of metallic hooks, ending in a spatula with beveled edges, that seems to allow a better pressure distribution on the skin and a deeper and more precise application, compared to the manual approach.

Recent studies indicate positive responses regrading pain intensity decrease in sports people suffering anterior knee pain, improving range of motion in subacromial impingement syndrome, improving sensory conductivity in symptomatic patients with carpal tunnel syndrome, decreased pain in patients with chronic epicondialgia or improveing function athletes with anterior knee pain.

However, the specific action mechanism, have not been investigated in depth yet. Clinical studies show improvements in strength, pain intensity, range of motion, or function. But whether if this effect is produced by changes in tissue tension or by reflexes effects, as has been suggested before, still unclear. There are no studies evaluating its effects on posterior muscular chain of lower extremity in athletes, where FD effects on neuromuscular response could be more evident due to the overload involved on this area.

Thus, the aim of this study is to evaluate the immediate, and after 30 minutes, effects of a single diacutaneous fibrolysis session on contractile and viscoelastic muscle properties and mechanosensitibity by means of tensiomyography, myotonometry and algometry on posterior muscular chain of lower limb in athletes.

DETAILED DESCRIPTION:
Diacutaneous fibrolysis is a physiotherapeutic instrumental technique, used to treat musculoskeletal conditions causing pain and/or movement restriction . It is applied by means of metallic hooks, ending in a spatula with beveled edges, that seems to allow a better pressure distribution on the skin and a deeper and more precise application, compared to the manual approach.

Recent studies indicate positive responses regrading pain intensity decrease in sports people suffering anterior knee pain, improving range of motion in subacromial impingement syndrome, improving sensory conductivity in symptomatic patients with carpal tunnel syndrome, decreased pain in patients with chronic epicondialgia or improveing function athletes with anterior knee pain.

However, the specific action mechanism, have not been investigated in depth yet. Clinical studies show improvements in strength, pain intensity, range of motion, or function. But whether if this effect is produced by changes in tissue tension or by reflexes effects, as has been suggested before, still unclear. There are no studies evaluating its effects on posterior muscular chain of lower extremity in athletes, where FD effects on neuromuscular response could be more evident due to the overload involved on this area.

Thus, the aim of this study is to evaluate the immediate, and after 30 minutes, effects of a single diacutaneous fibrolysis session on contractile and viscoelastic muscle properties and mechanosensitibity on posterior muscular chain of lower limb in athletes.

Design. A randomized controlled trial with blind evaluator. Randomization. Between lower extremities of each subject (Random.org). Regardless of its own dominance, diacutaneous fibrolysis will be applied to de following muscles and intermuscular septums: gluteus maixmus, biceps femoris and semitendinosus to de lower experimental limb. The other extremity will not be treat (control limb).

Sample recruitment. Athletes from UIC university community, who compete officially or institutionally, whether they are federated or recorded in a sport official register where the predominant activity focuses on the lower train (athletics, cycling, football, rugby...).

Procedure. The anthropometric data will be collected at the beginning of the study. The outcome assessment will be performed by a blinded evaluator at the baseline, immediately after the technique application and 30 minutes after.

An experienced physiotherapist in the diacutaneous fibrolysis technique will apply the treatment to the lower limb, previously randomized, in the following musculature and intermuscular septums: quadratus lumbar, gluteus maixum, biceps femoris and semitendinosus. Intervention procedure will last about 10-15 minutes

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign and have informed consent. They must have shortening of the hamstring muscles (being considered itself as such <160º in the Passive Knee Extension test as a main inclusion criteria.

Exclusion Criteria:

* Will involve any contraindication related to diacutaneous fibrolysis such us poor skin or trophic condition, taking anticoagulants, inflammatory process or recent injury).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-02-22 (Estimated); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-09-27 (Estimated)

PRIMARY OUTCOMES:
Contraction time changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Contraction time as a time between 10% and 90% of the contraction (ms). It will be assessed by tensomyography. Tensomyography is an evaluation method which allows to measure contractile muscle properties in isometric conditions, through an external electrical stimulus, of controlled intensity. It has a high of reliability (r = 0.93) and reproducibility.
  Tensomyography data for gluteus maximus, biceps femoris and semitendinosus, will be assessed, following protocols used in previous studies.
Relaxation time changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Relaxation time as a time between 90% and 50% of the relaxation (ms). It will be assessed by tensomyography. Tensomyography is an evaluation method which allows to measure contractile muscle properties in isometric conditions, through an external electrical stimulus, of controlled intensity. It has a high of reliability (r = 0.93) and reproducibility.
  Tensomyography data for gluteus maximus, biceps femoris and semitendinosus, will be assessed, following protocols used in previous studies.
Maximal Displacement changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Maximal displacement of the muscle contraction (mm). It will be assessed by tensomyography. Tensomyography is an evaluation method which allows to measure contractile muscle properties in isometric conditions, through an external electrical stimulus, of controlled intensity. It has a high of reliability (r = 0.93) and reproducibility.
  Tensomyography data for gluteus maximus, biceps femoris and semitendinosus, will be assessed, following protocols used in previous studies.
Contraction velocity changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Contraction velocity it is described as a change in Dm over time between 10% and 90% of the contraction (mm/s). It will be assessed by tensomyography. Tensomyography is an evaluation method which allows to measure contractile muscle properties in isometric conditions, through an external electrical stimulus, of controlled intensity. It has a high of reliability (r = 0.93) and reproducibility.
  Tensomyography data for gluteus maximus, biceps femoris and semitendinosus, will be assessed, following protocols used in previous studies.
Muscle tone changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Myotonometry is an assessing method for the viscoelastic characteristics of a resting muscle. It releases a mechanical impulse and provides quantitative values about muscle tone (Hz). This data will be collected at the same points used on tensiomyography .
  This data will be collected at the same points used on tensiomyography
Muscle Stiffness changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Muscle Stiffness changes will be assessed by myotonometry is an assessing method for the viscoelastic characteristics of a resting muscle. It releases a mechanical impulse and provides quantitative values about muscle stiffness (N/m). This data will be collected at the same points used on tensiomyography .
Mechanosensibility changes | at baseline, after diacutaneous fibrolysis intervention and 30 minutes later.
  Pressure algometry is a method that quantifies (Kg) mechanosensitivity, applying a mechanical stimulus of progressive compression on a point located in the body. In several studies, the trigger points, are the ones used for this purpose. Algometers are devices of easy accessibility, and is a method that has shown high reliability (r = 0.80) . This data will be collected at the same points used on tensomyography and myotonometry.
  This data will be collected at the same points used on tensiomyography

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cadellans-Arroniz A, Lopez-de-Celis C, Perez-Bellmunt A, Rodriguez-Sanz J, Llurda-Almuzara L, Gonzalez-Rueda V, Rodriguez-Rubio PR. Effects of Diacutaneous Fibrolysis on Passive Neuromuscular Response and Mechanosensitivity in Athletes with Hamstring Shortening: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jun 18;18(12):6554. doi: 10.3390/ijerph18126554. PMID 34207080